## Imperial College London

Hammersmith Hospital, Du Cane Road, London W12 0HS P: 02033133000 W: <a href="www.imperial.nhs.uk">www.imperial.nhs.uk</a>

Email: keenan.saleh10@imperial.ac.uk

Centre Number (if applicable):

Study Protocol Number: IRAS 330619
Patient Identification Number for this trial:

Full Title of Project: Unmasking Concealed Arrhythmia Syndromes

Name of Principal Investigator: Dr Zachary Whinnett

## Please initial box

| 1. | I confirm that I have read and understand the participant information sheet version dated for the above study and have had the opportunity to ask questions which have been answered fully. |
|---|---|
| 2. | I understand that my participation is voluntary, and I am free to withdraw at any time, without giving any reason and without my legal rights nor treatment / healthcare being affected. |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from Imperial College London, from NHS Trusts or from regulatory authorities where it is relevant to my taking part in this research. |
| 4. | I understand that data collected from me are a gift donated to Imperial College and that I will not personally benefit financially if this research leads to an invention and/or the successful development of a new test, medication treatment, product or service. |
| 5. | I give permission for my General Practitioner (GP) to be informed of my involvement in this study, and that any incidental findings of clinical significance will be communicated to them. |
| 6. | I consent to take part in the above study. |

## Please initial box

| | | Yes | No |
|---|---|---|---|
| | T | | |
| 7. | I give consent for information collected about me to be used to | | |
| | support other research or in the development of a new | | |
| | medical device or test by an academic institution or commercial company in the future, including those outside of | | |
| | the United Kingdom (which Imperial has ensured will keep this | | |
| | information secure). | | |
| 8. | I would like to be informed of the final anonymised results of | | |
| | the study via email. | | |

IRAS: 330619 Version 3 Date: 02/04/24



## Imperial College London

Hammersmith Hospital, Du Cane Road, London W12 0HS P: 02033133000 W: www.imperial.nhs.uk

| Email: keenan.saleh10@imper | ial.ac.uk |
|-----------------------------|-----------|
|-----------------------------|-----------|

| Name of Patient | Date | Signature |
|-------------------------------|------|-----------|
| Name of Person taking consent | Date | Signature |

1 copy for participant; 1 copy for Principal Investigator 1 copy for hospital notes

To ensure confidence in the process and minimise risk of loss, all consent forms must be printed, presented and stored in double sided format

IRAS: 330619 Version 3 Date: 02/04/24

